CLINICAL TRIAL: NCT02062658
Title: Extending Ketamine's Effects in Obsessive-Compulsive Disorder (OCD) With Exposure and Response Prevention (EX/RP)
Brief Title: Extending Ketamine's Effects in OCD With Exposure and Response Prevention (EX/RP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #6811; K23MH092434 (NIH)
Record Dates: First submitted 2014-02-12; First posted 2014-02-14 (Estimated); Results first posted 2016-10-27 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-11

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ketamine, Exposure & Response Prevention (Experimental): 0.5mg/kg IV Ketamine infusion followed by condensed course of Exposure and Response Prevention (EX/RP)
  Interventions: Drug: Ketamine; Behavioral: Exposure and Response Prevention

INTERVENTIONS:
Drug: Ketamine — 0.5mg/kg IV
  Other Names: Ketamine hydrochloride
Behavioral: Exposure and Response Prevention — A type of Cognitive Behavioral Therapy called Exposure and Response Prevention.
  Other Names: EX/RP

SUMMARY:
This study investigates if a single dose of IV Ketamine can rapidly improve Obsessive-Compulsive Disorder (OCD) symptoms and whether these effect can be maintained with a condensed course of a type of Cognitive Behavioral Therapy called Exposure and Response Prevention (EX/RP). You will be compensated for your time and travel. Participants must be between the ages of 18-55.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55
* Physically healthy and not currently pregnant
* Primary Diagnosis of OCD
* Sufficient severity of symptoms
* Currently off all psychotropic medication OR
* Currently on adequate dose of medication for treatment of OCD, but have not achieved at least partial remission
* Able to provide consent

Exclusion Criteria:

* Psychiatric conditions that make participation unsafe (schizophrenia [either self or first degree relative e.g. siblings, parents], history of violence, severe depression, eating disorder, substance dependence [including nicotine])
* Female patients who are either pregnant or nursing
* Planning to commence EX/RP during the period of the study or those who have completed an adequate dose of EX/RP (defined as 8 or more sessions within 2 months) within 8 weeks prior to enrollment.

period of the study

* Allergy to ketamine
* Participants for whom being off of medication is not clinically recommended
* Medical conditions that make participation unsafe (e.g. high blood pressure, head injury)
* Currently on medications that make participation unsafe

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H Blair Simpson, MD, PhD, Principal Investigator — Columbia-NYSPI-RFMH
Locations (1):
- New York State Psychiatric Insitute, New York, New York, United States

REFERENCES:
- [Result] Rodriguez CI, Wheaton M, Zwerling J, Steinman SA, Sonnenfeld D, Galfalvy H, Simpson HB. Can exposure-based CBT extend the effects of intravenous ketamine in obsessive-compulsive disorder? an open-label trial. J Clin Psychiatry. 2016 Mar;77(3):408-9. doi: 10.4088/JCP.15l10138. No abstract available. PMID 27046314

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult outpatients were recruited from the community starting March 2014 until March 2015.
Pre-assignment Details: No pre-assignment was done.
Period: Overall Study
Arm/Group | Ketamine, Exposure & Response Prevention
Started | 10
Completed | 8
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ketamine, Exposure & Response Prevention
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.3 (10.6)
Gender [Count of Participants; unit: Participants]
  Female | 1
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Met and Exceeded Response Criteria of Yale-Brown Obsessive-Compulsive Scale
Description: Patients given YBOCS (Yale Brown Obsessive-Compulsive Scale), a gold standard measure of obsessions and compulsions. For the YBOCS the minimum units are 0 and Maximum units on the total scale are 40. The higher the number on the YBOCS, the more severe the symptoms. Response was defined as at least a 35% reduction on the YBOCS.
Time Frame: 2 weeks
Measure: Number; unit: participants
Arm/Group | Ketamine, Exposure & Response Prevention
Number analyzed (Participants) | 8
participants | 5

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Ketamine, Exposure & Response Prevention
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No